CLINICAL TRIAL: NCT04053036
Title: Effects of MDMA on Responses to Affective Touch in Individuals With a Range of Autistic Traits
Brief Title: Effects of Drugs on Responses to Brain and Emotional Processes
Acronym: MAT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB19-0174
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-01

CONDITIONS: Autism Spectrum Disorder; Healthy
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Then MDMA (Experimental): Participants first receive placebo at their first session in the laboratory. Then will return to the laboratory 72 hours later and will receive MDMA (1.5 mg/kg)
  Interventions: Drug: MDMA; Drug: Placebo oral tablet
- MDMA Then Placebo (Experimental): Participants first receive MDMA (1.5 mg/kg) at their first session in the laboratory. Then will return to the laboratory 72 hours later and will receive placebo.
  Interventions: Drug: MDMA; Drug: Placebo oral tablet

INTERVENTIONS:
Drug: MDMA — Participants will be given 1.5mg/kg of MDMA
Drug: Placebo oral tablet — Participants will be given a placebo capsule that will only contain lactose.

SUMMARY:
To study the effects of a psychostimulant on responses to affective touch in individuals with a range of autistic traits

ELIGIBILITY:
Inclusion Criteria:

* BMI between 19 and 30 (no one under 130 lbs)
* Smokers smoking less than 25 cigarettes per week
* Have used ecstasy no more than 40 times with no adverse responses.

Exclusion Criteria:

* High blood pressure
* Any medical condition requiring regular medication
* Individuals with a current (within the last year) DSM-IV Axis 1 diagnosis
* Individuals with a history of dependence on stimulant drugs.
* Women who are pregnant or trying to become pregnant

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet de Wit, Principal Investigator — Principal Investigator
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Then MDMA | MDMA Then Placebo
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then MDMA | MDMA Then Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22
High School Education [Count of Participants; unit: Participants] | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Responses to Affective Touch
Description: Participants will complete an affective touch task during which time they will rate pleasantness of touch on a scale of -10 to +10 using an analog scale. Higher ratings indicate greater pleasantness.
Time Frame: 1.5 hrs after drug or placebo administration.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo oral tablet: Participants were given a placebo capsule that only contained lactose.
- MDMA: Participants first received MDMA (1.5 mg/kg) in a capsule
Arm/Group | Placebo | MDMA
Number analyzed (Participants) | 22 | 22
units on a scale | 3.01 (.7) | 4.06 (.5)

ADVERSE EVENTS:
Time Frame: .Through study completion, an average of 6 weeks.
Groups:
- Placebo: Placebo oral tablet: Participants will be given a placebo capsule that will only contain lactose.
Arm/Group | Placebo | MDMA
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/36/NCT04053036/Prot_SAP_000.pdf